CLINICAL TRIAL: NCT05767801
Title: Synovial Tissue and Blood Signature to Personalize the Management of Rheumatoid Arthritis Patients With Disease Flare After Biological DMARDs Discontinuation for Sustained Remission.
Brief Title: Synovial Tissue and Blood Signature of Rheumatoid Arthritis Patients With Disease Flare After Treatment Discontinuation for Sustained Remission.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Alivernini Stefano, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 2667
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Rheumatoid Arthritis
Keywords: synovial tissue; disease flare; sustained remission; peripheral blood
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RA patients in sustained clinical and ultrasound remission not changing treatment
  Interventions: Procedure: Evaluation of subclinical inflammation
- RA patients in sustained clinical and ultrasound remission changing treatment
  Interventions: Procedure: Evaluation of subclinical inflammation

INTERVENTIONS:
Procedure: Evaluation of subclinical inflammation — Minimally invasive synovial tissue biopsy for the semiquantitative and qualitative assessment of synovial immune and stromal cells; Peripheral blood collection for MBDA assessment and phenotyping of immune cells;

SUMMARY:
Flares of immune-mediated inflammatory diseases, as Rheumatoid Arthritis (RA), are a major burden for patients in routine care. They occur unpredictably, adding to the physical and psychological burden of the condition. In this study we will deeply dissect the synovial tissue and peripheral blood signature of RA in sustained remission eligible to treatment discontinuation to better understand the individualized factors determining disease flare once biological treatment is discontinued. We expect that the combined study of synovial tissue, imaging and peripheral blood derived biomarkers, associated with disease flare after treatment discontinuation in RA in remission, will provide a tool for the routine assessment of RA eligible to treatment discontinuation reducing the relapse rate and increasing the optimization of the use of expensive pharmacological treatments only for patients still needing them.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of RA following the 2010 ACR/EULAR classification criteria
* Age ≥18 and ≤75 years
* Sustained remission (DAS<1.6 for at least 3 sequential evaluations 6months apart).
* Without evidence of ultrasound detected synovitis (Power Doppler negative in knee, wrist, II-V MCP, II-V PIP and II-V MTP bilaterally).
* Patients under treatment with stable dose of conventional, synthetic or biological DMARDs.
* Patients without steroid treatment in the last 6 months.

Exclusion Criteria:

* With other diagnosis of chronic joint diseases rather than RA.
* Unable to participate to the clinical outpatient follow-up.
* Exposed to steroid treatment within 6 months from study screening.
* With evidence of ultrasound detected synovitis (Power Doppler positivity) in other joints than the ones included in the screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Rheumatoid Arthritis in stable remission (DAS<1.6 for at least 6 months) and under treatment with stable dose of conventional, synthetic or biological DMARDs. All patients at the time of enrolment must fulfil the ultrasound criteria of Power Doppler negativity of knee, wrist, II-V MCP and II-V MTP bilaterally and any other reported painful joint not included in the screening ultrasound protocol.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2023-03-14 (Estimated)

PRIMARY OUTCOMES:
Disease flare rate | 24 months

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - UOC Reumatologia - Policlinico di Bari, Bari, Apulia
  - Centro di Ricerca E. Menni - Fondazione Poliambulanza Brescia, Brescia, Lombardy
  - Division of Rheumatology, Rome

IPD SHARING:
Plan to Share IPD: No